CLINICAL TRIAL: NCT04627935
Title: The Effect of Foot Deformities on Physical Activity, Fatigue Level and Quality of Life in Elderly COPD Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2020.766
Record Dates: First submitted 2020-11-08; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Chronic Obstructive Pulmonary Disease; Foot Deformities; Quality of Life; Activity, Motor; Fatigue
Keywords: Chronic Obstructive Pulmonary Disease; Foot deformities; quality of life; physical activity; fatigue; geriatric patient
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Foot Deformities; Motor Activity; Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD patients: Patients with a diagnosis of COPD aged over 60 years
  Interventions: Behavioral: The COPD Assessment Test; Diagnostic Test: Navicular Drop Test; Behavioral: International Physical Activity Questionnaires (IPAQ); Behavioral: COPD and Asthma Fatigue Scale (CAFS); Behavioral: Saint George Respiratory Questionnaire

INTERVENTIONS:
Behavioral: The COPD Assessment Test — Used to assess symptoms in COPD patients.
Diagnostic Test: Navicular Drop Test — It is the test used to measure the amount of pronation in the foot.
Behavioral: International Physical Activity Questionnaires (IPAQ) — The International Physical Activity Questionnaires (IPAQ) comprises a set of 4 questionnaires. The purpose of the questionnaires is to provide common instruments that can be used to obtain internationally comparable data on health-related physical activity.
Behavioral: COPD and Asthma Fatigue Scale (CAFS) — CAFS is a comprehensive, brief, patient-centered questionnaire developed to capture fatigue experienced by patients with asthma or COPD.
Behavioral: Saint George Respiratory Questionnaire — Disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease.

SUMMARY:
The aim of this study is to investigate the effects of changes in foot structure on physical activity level, fatigue and quality of life in COPD patients.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is usually a progressive disease associated with the increased chronic inflammatory response of the airways and lungs to the toxic effects of harmful gases and particles. It causes pathological changes such as increased secretion production in the airways, epithelial changes, inflammation, smooth muscle hypertrophy, and hyperplasia in the submucosal glands. Hyperinflammation in the lungs results in muscle atrophy, shortening of the respiratory muscles, and increased respiratory workload. On the other hand, the increase in pro-inflammatory plasma cytokine levels seen in the systemic circulation causes oxidative stress, leading to the development of musculoskeletal system disorders and a decrease in functional capacity. Pulmonary dysfunction and increased dyspnea lead to a decrease in physical condition, physical exercise tolerance, and activity, while the decrease in muscle mass results in atrophy in the peripheral extremities.

Age and gender are cited as major risk factors for COPD. Therefore, lower extremity atrophy, which is seen in peripheral extremities and increases with aging, causes foot dysfunctions. Considering that the ability of elderly people to maintain their independence is related to a good level of consciousness and ongoing ambulation, and the frequency of foot problems seen in elderly people is approximately twice as high as the general population, foot problems seen in elderly individuals are very important for this group. In particular, the decrease in foot mobility and the fall of the medial longitudinal arch negatively affect the absorption of shocks during heel strike and foot flat and the momentum of the trunk forward. This situation may result in the expenditure of energy above normal and deterioration of balance while ensuring the proper transfer of body weight. All of these cause early fatigue and a decrease in the quality of life in the individual. In the literature, foot deformities in elderly healthy individuals and the parameters these deformities will affect people are stated. However, there is no study examining the effects of foot deformities on physical activity, fatigue, and quality of life in elderly COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of COPD
* Age over 60

Exclusion Criteria:

* Having an orthopedic or neurological disorder that affects the walking pattern
* Having a peripheral vascular disease
* Being diagnosed with Diabetes Mellitus
* Having systemic diseases such as arthritis
* Having a previous history of foot-ankle fractures
* Having a dermatological disease (fungal and bacterial infection etc.)

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 77 COPD patients, over 60 years of age
Sampling Method: Non-Probability Sample
Enrollment: 77 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Navicular Drop Test | Day 0
  It is the test used to measure the amount of pronation in the foot.

SECONDARY OUTCOMES:
The COPD Assessment Test | Day 0
  Used to assess symptoms in COPD patients.
International Physical Activity Questionnaires (IPAQ) | Day 0
  The International Physical Activity Questionnaires (IPAQ) comprises a set of 4 questionnaires. The purpose of the questionnaires is to provide common instruments that can be used to obtain internationally comparable data on health-related physical activity.
COPD and Asthma Fatigue Scale (CAFS) | Day 0
  CAFS is a comprehensive, brief, patient-centered questionnaire developed to capture fatigue experienced by patients with asthma or COPD.
Saint George Respiratory Questionnaire | Day 0
  Disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease.

CONTACTS AND LOCATIONS:
Overall Officials: Nilufer Kablan, Asst. Prof., Study Director — Istanbul Sağlık Bilimleri University; Ayca Evkaya Acar, Res. Asst., Principal Investigator — Maltepe University
Locations (1):
- Istanbul Saglık Bilimleri University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Jones PW, Adamek L, Nadeau G, Banik N. Comparisons of health status scores with MRC grades in COPD: implications for the GOLD 2011 classification. Eur Respir J. 2013 Sep;42(3):647-54. doi: 10.1183/09031936.00125612. Epub 2012 Dec 20. PMID 23258783
- [Background] de Sa RB, Pessoa MF, Cavalcanti AGL, Campos SL, Amorim C, Dornelas de Andrade A. Immediate effects of respiratory muscle stretching on chest wall kinematics and electromyography in COPD patients. Respir Physiol Neurobiol. 2017 Aug;242:1-7. doi: 10.1016/j.resp.2017.03.002. Epub 2017 Mar 10. PMID 28286249
- [Background] Sun KS, Lin MS, Chen YJ, Chen YY, Chen SC, Chen W. Is asymptomatic peripheral arterial disease associated with walking endurance in patients with COPD? Int J Chron Obstruct Pulmon Dis. 2015 Jul 29;10:1487-92. doi: 10.2147/COPD.S85430. eCollection 2015. PMID 26251588
- [Background] Atasever A, Erdinc E. [Quality of life in COPD]. Tuberk Toraks. 2003;51(4):446-55. Turkish. PMID 15143396
- [Background] Theander K, Unosson M. Fatigue in patients with chronic obstructive pulmonary disease. J Adv Nurs. 2004 Jan;45(2):172-7. doi: 10.1046/j.1365-2648.2003.02878.x. PMID 14706002